CLINICAL TRIAL: NCT05121350
Title: A Multicenter, Randomized, Double-blind, Parallel-controlled Phase III Trial to Evaluate the Efficacy and Safety of Anotinib Hydrochloride Capsule Combined With Epirubicin Hydrochloride Versus Placebo Combined With Epirubicin Hydrochloride in First-line Treatment of Advanced Soft Tissue Sarcoma
Brief Title: A Clinical Trial to Evaluate the Efficacy and Safety of Anotinib Hydrochloride Capsule Combined With Epirubicin Hydrochloride Versus Placebo Combined With Epirubicin Hydrochloride in First-line Treatment of Advanced Soft Tissue Sarcoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALTN-III-04
Record Dates: First submitted 2021-11-15; First posted 2021-11-16 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Epirubicin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arotinib hydrochloride capsule + Epirubicin (Experimental): Arotinib hydrochloride capsule combined with epirubicin, 21 days as a treatment cycle
  Interventions: Drug: Anlotinib hydrochloride capsule; Drug: Epirubicin
- Placebo + Epirubicin (Active Comparator): Placebo combined with epirubicin, 21 days as a treatment cycle
  Interventions: Drug: Epirubicin; Drug: Arotinib hydrochloride capsule placebo

INTERVENTIONS:
Drug: Anlotinib hydrochloride capsule — Anlotinib hydrochloride is a multi-target tyrosine kinase inhibitor.
  Arms: Arotinib hydrochloride capsule + Epirubicin
Drug: Epirubicin — Epirubicin can inhibit the synthesis of DNA and RNA.
Drug: Arotinib hydrochloride capsule placebo — Placebo of Anlotinib hydrochloride capsule
  Arms: Placebo + Epirubicin

SUMMARY:
A multicenter, randomized, double-blind, parallel-controlled Phase III trial to evaluate the efficacy and safety of anotinib hydrochloride capsule combined with epirubicin hydrochloride versus placebo combined with epirubicin hydrochloride in first-line treatment of advanced soft tissue sarcoma

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1.
* Life expectancy >=3 months.
* Female patients of childbearing age should agree to use contraceptive measures during the study period and for at least 6 months after study is stopped; male patients should agree to use contraception during the study period and for at least 6 months after study is stopped.
* Understood and signed an informed consent form.

Exclusion Criteria:

* Diagnosed and/or treated additional malignancy within 5 years before the first dose.
* With factors affecting oral medication.
* Received major surgical treatment, open biopsy or obvious traumatic injury within 4 weeks before the first dose.
* A history of psychotropic drug abuse or have a mental disorder.
* Any severe and/or uncontrolled diseas.
* Has received Chinese patent medicines with anti-tumor indications within 2 weeks before the first dose.
* Has participated in other clinical studies within 4 weeks before the first dose.
* According to the judgement of the investigators, there are other factors that subjects are not suitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) assessed by independent review committees (IRC) | Baseline up to 12 months
  Time from the first dose to the first documentation of progression disease (PD) or death from any cause, whichever occurs first

SECONDARY OUTCOMES:
Overall survival (OS) | Baseline up to die
  From randomization to the time of death from any cause
progression free survival (PFS) assessed by investigator | Baseline up to 12 months
  Time from the first dose to the first documentation of PD or death from any cause, whichever occurs first
Objective response rate (ORR) | Baseline up to 6 months
  The sum of percentage of participants with complete response rate and partial response rate
Disease control rate (DCR) | Baseline up to 25 months
  percentage of participants with complete response, partial response plus stable disease
Duration of overall response (DOR) | Baseline up to 6 months
  the time from the date of first documentation of a CR or PR to the date of first documentation of tumor progression
Degradation rate | Baseline up to 6 months
  Proportion of patients with tumor regression meeting surgical resection criteria in each group during the study period

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Beijing Jishuitan Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Fudan University Zhongshan Hospital, Shanghai, Shanghai Municipality